CLINICAL TRIAL: NCT04827485
Title: Gluteal Squeeze for Left Colon Distension During Withdrawal in Colonoscopy
Brief Title: Gluteal Squeeze for Left Colon Distension
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decision.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Douglas K. Rex, Professor Emeritus, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: 11109
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gluteal squeeze (Active Comparator): Patients behind pressed together during part of the colonoscopy (The technicians arms will be covered with a towel to mask the provider of any pressure being applied)
  Interventions: Other: Gluteal squeeze
- Non-squeeze (Sham Comparator): When the doctor asks for gluteal pressure, a technician will not administer the pressure but their arms will be covered with a towel and the doctor will not know if the pressure is being administered or not.
  Interventions: Other: No squeeze

INTERVENTIONS:
Other: Gluteal squeeze — During procedure, the doctor performing colonoscopy will ask for gluteal pressure. The technician will perform the maneuver, but the doctor will be blinded as the arms of the technician along with the patients behind are covered by a towel.
  Arms: Gluteal squeeze
Other: No squeeze — During procedure, the doctor performing colonoscopy will ask for gluteal pressure. The technician will not perform the maneuver, but the doctor will be blinded as the arms of the technician along with the patients behind are covered by a towel.
  Arms: Non-squeeze

SUMMARY:
Good distension of the colon during colonoscopy is essential to detect polyps. Gas sometimes escapes the colon through the anus resulting in compromised distension. Pressure on gluteal muscles when the colonoscope tip is in the left colon might help preventing this and thus increase visibility. No previous study looked at this.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 40 years
2. Scheduled colonoscopy

Exclusion Criteria:

1. Inflammatory bowel disease
2. History of colorectal cancer or colon resection
3. Any colorectal cancer syndromes (FAP, HNPCC, SPS)
4. Patient with poor bowel preparation identified during insertion

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Left colon distension score | during the procedure
  Provider reported distension score in the left colon

SECONDARY OUTCOMES:
Left colon withdrawal time | during the procedure
  Time taken to withdraw the scope in the left colon
Left colon examination time | during the procedure
  Time taken to inspect during left colon withdrawal
Left colon adenoma detection rate | during the procedure
  proportion of patients with at least one left colon adenoma
Left colon sessile serrated lesion detection rate | during the procedure
  proportion of patients with at least one left colon sessile serrated lesion

CONTACTS AND LOCATIONS:
Overall Officials: Douglas K Rex, MD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - IU Health University Hospital, Indianapolis, Indiana
  - Spring Mill Medical Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaminski MF, Wieszczy P, Rupinski M, Wojciechowska U, Didkowska J, Kraszewska E, Kobiela J, Franczyk R, Rupinska M, Kocot B, Chaber-Ciopinska A, Pachlewski J, Polkowski M, Regula J. Increased Rate of Adenoma Detection Associates With Reduced Risk of Colorectal Cancer and Death. Gastroenterology. 2017 Jul;153(1):98-105. doi: 10.1053/j.gastro.2017.04.006. Epub 2017 Apr 17. PMID 28428142
- [Background] Corley DA, Jensen CD, Marks AR, Zhao WK, Lee JK, Doubeni CA, Zauber AG, de Boer J, Fireman BH, Schottinger JE, Quinn VP, Ghai NR, Levin TR, Quesenberry CP. Adenoma detection rate and risk of colorectal cancer and death. N Engl J Med. 2014 Apr 3;370(14):1298-306. doi: 10.1056/NEJMoa1309086. PMID 24693890
- [Background] Rex DK, Schoenfeld PS, Cohen J, Pike IM, Adler DG, Fennerty MB, Lieb JG 2nd, Park WG, Rizk MK, Sawhney MS, Shaheen NJ, Wani S, Weinberg DS. Quality indicators for colonoscopy. Am J Gastroenterol. 2015 Jan;110(1):72-90. doi: 10.1038/ajg.2014.385. Epub 2014 Dec 2. No abstract available. PMID 25448873
- [Background] Rex DK. Colonoscopic withdrawal technique is associated with adenoma miss rates. Gastrointest Endosc. 2000 Jan;51(1):33-6. doi: 10.1016/s0016-5107(00)70383-x. PMID 10625792
- [Background] Woltjen JA. A retrospective analysis of cecal barotrauma caused by colonoscope air flow and pressure. Gastrointest Endosc. 2005 Jan;61(1):37-45. doi: 10.1016/s0016-5107(04)02453-8. PMID 15672054
- [Background] Duloy A, Yadlapati RH, Benson M, Gawron AJ, Kahi CJ, Kaltenbach TR, McClure J, Gregory DL, Keswani RN. Video-Based Assessments of Colonoscopy Inspection Quality Correlate With Quality Metrics and Highlight Areas for Improvement. Clin Gastroenterol Hepatol. 2019 Mar;17(4):691-700. doi: 10.1016/j.cgh.2018.05.060. Epub 2018 Jun 14. PMID 29908363